CLINICAL TRIAL: NCT06925542
Title: A Phase 1 Dose Evaluation Study of the Safety and Preliminary Efficacy of Anti-CD19 Allogeneic CRISPR-Cas9-Engineered T Cells (CTX112) in Adult Subjects With Refractory Autoimmune Disease
Brief Title: A Safety and Efficacy Study Evaluating CTX112 in Adult Subjects With Refractory Autoimmune Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-AID-500
Record Dates: First submitted 2025-03-25; First posted 2025-04-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: SLE (Systemic Lupus); Lupus Erythematosus, Systemic; Lupus Nephritis; Systemic Sclerosis; Inflammatory Myopathy, Idiopathic; Myositis; Diffuse Cutaneous Systemic Sclerosis
Keywords: CAR T; Lupus; SLE; Lupus Nephritis; Allogeneic; CD19; Cell Therapy; Scleroderma; Myositis; Systemic sclerosis; Idiopathic Inflammatory Myopathy; Inflammatory Myopathy; Diffused Cutaneous Systemic Sclerosis; Gene Therapy; Autoimmune
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Scleroderma, Systemic; Myositis; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX112 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy
  Interventions: Biological: CTX112

INTERVENTIONS:
Biological: CTX112 — CTX112 (CD19-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components)

SUMMARY:
This is a single-arm, open-label, multicenter, ascending dose Phase 1 study evaluating the safety and preliminary efficacy of CTX112 in adult subjects with refractory autoimmune diseases, including active systemic lupus erythematosus (SLE), systemic sclerosis (SSc), or idiopathic inflammatory myopathy (IIM).

DETAILED DESCRIPTION:
This study may enroll up to 80 subjects in total. CTX112 is a CD19 directed chimeric antigen receptor (CAR) T cell immunotherapy comprised of allogeneic T cells prepared for the treatment of refractory autoimmune diseases. The cells are from healthy adult volunteer donors that are genetically modified ex vivo using CRISPR-Cas9 (clustered regularly interspaced short palindromic repeats/ CRISPR-associated protein 9) gene editing components (single guide RNA and Cas9 nuclease).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years and < 70 years of age.
2. Subjects must voluntarily sign a written informed consent and be willing and able to comply with all study requirements.
3. Adequate hematologic, renal, liver, cardiac and pulmonary organ function.
4. Subjects must agree to use acceptable methods of contraception.
5. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, contraceptive guidelines, and other study procedures.
6. Diagnosis of systemic lupus erythematosus (SLE), systemic sclerosis (SSc) or idiopathic inflammatory myopathy (IIM).

For systemic lupus erythematosus (SLE) subjects:

- Diagnosis of SLE by a board-certified rheumatologist that conforms with 2019 ACR/EULAR criteria. For lupus nephritis subjects, active, biopsy-proven proliferative lupus nephritis Class III or IV, either with or without the presence of Class V, and appropriate National Institutes of Health index activity score using the 2018 International Society of Nephrology/Renal Pathology Society criteria.

For Systemic Sclerosis (SSc) subjects:

- Diagnosis of diffuse cutaneous systemic sclerosis (dcSSC) or SSc-ILD that conforms with 2013 ACR/EULAR criteria. Subjects should meet active skin or lung disease criteria.

For Idiopathic Inflammatory Myopathy (IIM) subjects:

- Diagnosis with dermatomyositis (DM), polymyositis (PM) or myositis as part of rheumatologic overlap syndrome, antisynthetase (ASyS), or immune-mediated necrotizing myopathy (IMNM) that conforms with 2017 ACR/EULAR criteria for inflammatory myopathies. Subjects must meet moderate severe, skin, or lung involvement criteria.

Key Exclusion Criteria:

1. Prior anti-CD19 therapy or any gene therapy/genetically modified cell therapy.
2. Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant.
3. Severe active or history of central nervous (CNS) involvement.
4. History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease or any autoimmune disease with CNS involvement other than SLE, SSc or IIM.
5. Mixed connective tissue disease with no clear predominant disease.
6. Presence of study disease manifestations or other conditions that are likely to pose increase safety risks and/or confound disease assessments, or pose significant risk to those receiving CAR T cell therapy.
7. History of primary or secondary immunodeficiency.
8. Presence or history of certain bacterial, viral or fungal infection.
9. Malignancy in the last 5 years (with the exception of cancers deemed to be low likelihood for recurrence).
10. Diagnosis of a genetic disorder associated with bone marrow failure or myelodysplastic syndrome.
11. History or current diagnosis of catastrophic anti-phospholipid syndrome or anti phospholipid syndrome that requires ongoing anticoagulation.
12. Pregnant or lactating.
13. Presence or history of disease requiring treatment that is not compatible with the study protocol; presence or history of other conditions that are not compatible with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CTX112 in adult subjects with refractory autoimmune diseases, including SLE, SSc or IIM | From CTX112 infusion up to 28 days post-infusion
  Incidence of dose-limiting toxicities

SECONDARY OUTCOMES:
To assess the pharmacodynamic response of CTX112 in adult subjects with refractory autoimmune diseases, including SLE, SSc or IIM | From CTX112 infusion up to 60 months post-infusion
  Change from baseline in disease specific autoantibody markers
To assess the pharmacokinetics (PK) of CTX112 in adult subjects with refractory autoimmune diseases, including SLE, SSc or IIM | From CTX112 infusion up to 60 months post-infusion
  Levels of CTX112 in blood over time
To assess the preliminary efficacy of CTX112 in adult subjects with refractory autoimmune diseases, including active SLE, SSc or IIM. | From CTX112 infusion up to 60 months post-infusion
  For SLE subjects: disease response rates based on SLEDAI-2K instrument; DORIS and LLDAS criteria
  For SSc subjects: disease response rates based on ACR-CRISS (including mRSS, forced vital capacity, HAQ-DI, Physician Global Assessment, Patient Global Assessment)
  For IIM subjects: disease response rates based on ACR/EULAR total Improvement score (including MMT8, EMDA, forced vital capacity, Physician Global Assessment, Patient Global Assessment, muscle enzyme level)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Research Site 4, Redwood City, California
  - Research Site 2, Chicago, Illinois
  - Research Site 8, Iowa City, Iowa
  - Research Site 6, Boston, Massachusetts
  - Research Site 1, St Louis, Missouri
  - Research Site 5, Chapel Hill, North Carolina
- Germany (2):
  - Research Site 7, Augsburg
  - Research Site 3, Hanover

IPD SHARING:
Plan to Share IPD: No